CLINICAL TRIAL: NCT04096742
Title: A Prospective, Randomized, Double-blind, Vehicle-controlled Study Evaluating the Efficacy, Safety and Patient Satisfaction of Tretinoin 0.05% Lotion (Altreno) for Chest Rejuvenation.
Brief Title: Altreno for Chest Rejuvenation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Altreno-2019-01
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Photodamaged Skin; Photoaging
Keywords: Skin; Chest; Photodamage; Sun Damage
MeSH Terms: interventions — Tretinoin

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, double-blind, randomized, vehicle-controlled study
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Altreno (Experimental): tretinoin 0.05% lotion (Altreno)
  Interventions: Drug: tretinoin 0.05% lotion (Altreno)
- Vehicle (Sham Comparator): Vehicle lotion not containing tretinoin
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: tretinoin 0.05% lotion (Altreno) — Altreno topical lotion
  Arms: Altreno
Other: Vehicle — Lotion not containing active ingredient (tretinoin)
  Arms: Vehicle

SUMMARY:
This is a single-center, prospective, double-blind, randomized, vehicle-controlled study to evaluate the efficacy, safety and patient satisfaction of tretinoin 0.05% lotion (Altreno) for chest rejuvenation.

ELIGIBILITY:
Inclusion Criteria:

1. Females or males age 18-65, Fitzpatrick skin types I-VI
2. Moderate to severe photodamage (Fitzpatrick Wrinkle score of 4-9)
3. Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedures.
4. Willingness to abstain from any other procedures to the areas to be treated throughout the trial period.
5. Willingness and ability to comply with protocol requirements, including adherence to photography and returning for follow-up visits.
6. Women of childbearing potential willing to use an acceptable form of birth control during trial period.

   1. Hormonal contraception - pill, injection, implant, patch, vaginal ring, Intrauterine device
   2. Intrauterine coil
   3. Barrier method used with an additional form of contraception (e.g., sponge, spermicide or condom)
   4. Abstinence (If practicing abstinence must agree to use barrier method described above (c) if becomes sexually active).
   5. Vasectomized partner (Must agree to use barrier method described above (c) if becomes sexually active with an Un-Vasectomized partner).
7. Female patients will be either of non-childbearing potential defined as: Having no uterus and/or both ovaries, postmenopausal (no menses for at least 12 months prior), or has had a bilateral tubal ligation at least 6 months prior to study enrollment.

Exclusion Criteria:

1. Pregnancy, currently breast feeding or planning pregnancy for the duration of the trial.
2. Known hypersensitivity or allergy to the components of the study medication.
3. Concurrent enrollment in any study involving the use of investigational devices or drugs.
4. Current smoker or history of smoking in the last five years.
5. Current user of any nicotine-containing products, e.g., e-cigarettes, Nicorette gum, nicotine patches, etc.
6. Presence of an active systemic or local skin disease that may affect treatment area.
7. History of prior surgery to the treatment area
8. History of prior significant trauma to the chest
9. History of the following cosmetic treatments to the area(s) to be treated:

   1. Energy based device or laser procedure to the chest within the past 6 months (Ultherapy, ablative and non-ablative laser, intense pulsed light, etc)
   2. Injectable filler of any type to the chest in the past 2 years (Hyaluronic acid fillers (Voluma, Belotero), Poly-L-Lactic acid fillers (e.g. Sculptra), and CaHA fillers (e.g. Radiesse)
   3. Ever for permanent fillers (e.g. Silicone, ArteFill)
10. Surgical dermabrasion or chemical peels in the treatment area within the past 6 month
11. Any planned surgical intervention to the chest for the duration of the trial
12. Any visible surface alteration to the chest that may interfere with evaluation, at investigator discretion
13. Any pre-existing medical condition that may interfere with study compliance or evaluation, at investigator discretion
14. Inability to comply with all study protocols and regulations
15. Current taking an immunosuppressant or applying a topical corticosteroid to the affected area
16. Unwilling to minimize exposure to sunlight and sunlamps during the course of the study.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-06 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Skin Quality | Baseline through Month 6
  Nine-point scale to assess skin quality for the appearance of crepiness, coarse lines/wrinkles, skin texture, and skin tone evenness

SECONDARY OUTCOMES:
Investigator Assessment-Fabi-Bolton Wrinkle Scale (FBWS) | Baseline through Month 6
  Fabi-Bolton Wrinkle Scale (FBWS)
Investigator Assessment-Investigator Percent Improvement Evaluation | 1, 3, and 6 months
  Investigator Percent Improvement Evaluation
Investigator Assessment-Investigator Global aesthetic improvement scale (I-GAIS) | 1, 3, and 6 months
  Investigator Global aesthetic improvement scale (I-GAIS)
Subject Assessments-Subject Global aesthetic improvement scale (S-GAIS) | 1, 3, and 6 months
  Subject Global aesthetic improvement scale (S-GAIS)
Subject Assessments-Patient satisfaction score | 1, 3, and 6 months
  Patient satisfaction score
Subject Assessments-End of study patient questionnaire | Month 6
  End of study patient questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Fabi, MD, Principal Investigator — Cosmetic Laser Dermatology
Locations (1):
- Cosmetic Laser Dermatology/West Dermatology Research Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No